CLINICAL TRIAL: NCT01773967
Title: Impact of Emergency Department Probiotic (LGG) Treatment of Pediatric Gastroenteritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Columbia University (Other); Northwestern University (Other); University of New Mexico (Other); Children's National Research Institute (Other); University of Utah (Other); Wayne State University (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Michigan (Other); Brown University (Other); University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01HD071915 (NIH); NCT00970164 (obsolete NCT alias)
Record Dates: First submitted 2013-01-10; First posted 2013-01-23 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Gastroenteritis
Keywords: Lactobacillus rhamnosus GG; LGG; Probiotic; Gastroenteritis; acute gastroenteritis; child; pediatric; RCT
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LGG (Experimental): LGG 10^10 cfu PO bid x 5 days
  Interventions: Drug: LGG
- Placebo (Placebo Comparator): micro-crystalline cellulose PO bid x 5 days
  Interventions: Drug: micro-crystalline cellulose

INTERVENTIONS:
Drug: LGG — LGG 10^10 cfu PO BID X 5 days
  Other Names: Lactobacillus GG ATCC 53103; Lactobacillus rhamnosus; culturelle
  Arms: LGG
Drug: micro-crystalline cellulose — 1 capsule PO bid x 5 days
  Other Names: placebo micro-crystalline cellulose
  Arms: Placebo

SUMMARY:
The investigators will study the efficacy and side effect profile of LGG, a probiotic, in pediatric patients with acute gastroenteritis.

DETAILED DESCRIPTION:
Multicenter randomized controlled trial of LGG in patients 3-48 months of age presenting to the Emergency Department with acute gastroenteritis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-48 months (have not yet reached their fourth birthday); AND
2. Presence of 3 or more watery stools within 24 hours of screening; AND
3. Duration of vomiting or diarrhea less than 7 days; AND
4. Symptoms consistent with acute intestinal infectious process.

Exclusion Criteria:

1. Presence of an indwelling vascular access line; OR
2. Presence of structural heart disease excluding non-pathological heart murmurs; OR
3. Receiving immunosuppressive therapy or history of immunodeficiency; OR
4. Hematochezia in the preceding 48 hours; OR
5. Chronic gastrointestinal problems (e.g. short gut syndrome, inflammatory bowel disease); OR
6. Patients with known pancreatitis; OR
7. History of abdominal surgery; OR
8. Critically ill patients; OR
9. Family member with an indwelling vascular access line, or on immunosuppressive therapy, or with a known immunodeficiency; OR
10. Bilious emesis; OR
11. Probiotic use (supplement) in the preceding 2 weeks; OR
12. Oral or intravenous steroid use in the preceding six months; OR
13. Previously enrolled in this trial; OR
14. Allergy to lactobacillus or Microcrystalline Cellulose (MCC); OR
15. Allergy to erythromycin, clindamycin, AND betalactam antibiotics (all); OR
16. Not available for daily follow-up while symptomatic; OR
17. Parent/guardian not speaking English or Spanish; OR
18. Under 6 months old AND premature (<37 weeks).

Ages: 3 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 971 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Quayle, MD, Principal Investigator — Washington University School of Medicine
Locations (10):
- United States (10):
  - UC Davis Medical Center, Sacramento, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital, Chicago, Illinois
  - University of Michigan Health System, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - Children's Hospital of New York, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Hasbro Children's Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Freedman SB, Finkelstein Y, Pang XL, Chui L, Tarr PI, VanBuren JM, Olsen C, Lee BE, Hall-Moore CA, Sapien R, O'Connell K, Levine AC, Poonai N, Roskind C, Schuh S, Rogers A, Bhatt S, Gouin S, Mahajan P, Vance C, Hurley K, Powell EC, Farion KJ, Schnadower D. Pathogen-Specific Effects of Probiotics in Children With Acute Gastroenteritis Seeking Emergency Care: A Randomized Trial. Clin Infect Dis. 2022 Aug 24;75(1):55-64. doi: 10.1093/cid/ciab876. PMID 34596225
- [Derived] Schnadower D, O'Connell KJ, VanBuren JM, Vance C, Tarr PI, Schuh S, Hurley K, Rogers AJ, Poonai N, Roskind CG, Bhatt SR, Gouin S, Mahajan P, Olsen CS, Powell EC, Farion K, Sapien RE, Chun TH, Freedman SB; Pediatric Emergency Care Applied Research Network and Pediatric Emergency Research Canada. Association Between Diarrhea Duration and Severity and Probiotic Efficacy in Children With Acute Gastroenteritis. Am J Gastroenterol. 2021 Jul 1;116(7):1523-1532. doi: 10.14309/ajg.0000000000001295. PMID 34183579
- [Derived] Freedman SB, Roskind CG, Schuh S, VanBuren JM, Norris JG, Tarr PI, Hurley K, Levine AC, Rogers A, Bhatt S, Gouin S, Mahajan P, Vance C, Powell EC, Farion KJ, Sapien R, O'Connell K, Poonai N, Schnadower D; Pediatric Emergency Research Canada and Pediatric Emergency Care Applied Research Networks. Comparing Pediatric Gastroenteritis Emergency Department Care in Canada and the United States. Pediatrics. 2021 Jun;147(6):e2020030890. doi: 10.1542/peds.2020-030890. Epub 2021 May 20. PMID 34016656
- [Derived] Poonai N, Powell EC, Schnadower D, Casper TC, Roskind CG, Olsen CS, Tarr PI, Mahajan P, Rogers AJ, Schuh S, Hurley KF, Gouin S, Vance C, Farion KJ, Sapien RE, O'Connell KJ, Levine AC, Bhatt S, Freedman SB; Pediatric Emergency Care Applied Research Network (PECARN) and Pediatric Emergency Research Canada (PERC). Variables Associated With Intravenous Rehydration and Hospitalization in Children With Acute Gastroenteritis: A Secondary Analysis of 2 Randomized Clinical Trials. JAMA Netw Open. 2021 Apr 1;4(4):e216433. doi: 10.1001/jamanetworkopen.2021.6433. PMID 33871616
- [Derived] Schnadower D, Sapien RE, Casper TC, Vance C, Tarr PI, O'Connell KJ, Levine AC, Roskind CG, Rogers AJ, Bhatt SR, Mahajan P, Powell EC, Olsen CS, Gorelick MH, Dean JM, Freedman SB; Pediatric Emergency Care Applied Research Network (PECARN) Probiotics Study. Association between Age, Weight, and Dose and Clinical Response to Probiotics in Children with Acute Gastroenteritis. J Nutr. 2021 Jan 4;151(1):65-72. doi: 10.1093/jn/nxaa313. PMID 33274370
- [Derived] Schnadower D, Tarr PI, Casper TC, Gorelick MH, Dean JM, O'Connell KJ, Mahajan P, Levine AC, Bhatt SR, Roskind CG, Powell EC, Rogers AJ, Vance C, Sapien RE, Olsen CS, Metheney M, Dickey VP, Hall-Moore C, Freedman SB. Lactobacillus rhamnosus GG versus Placebo for Acute Gastroenteritis in Children. N Engl J Med. 2018 Nov 22;379(21):2002-2014. doi: 10.1056/NEJMoa1802598. PMID 30462938
- [Derived] Schnadower D, Tarr PI, Casper TC, Gorelick MH, Dean MJ, O'Connell KJ, Mahajan P, Chun TH, Bhatt SR, Roskind CG, Powell EC, Rogers AJ, Vance C, Sapien RE, Gao F, Freedman SB. Randomised controlled trial of Lactobacillus rhamnosus (LGG) versus placebo in children presenting to the emergency department with acute gastroenteritis: the PECARN probiotic study protocol. BMJ Open. 2017 Sep 24;7(9):e018115. doi: 10.1136/bmjopen-2017-018115. PMID 28947466
- [Derived] Freedman SB, Williamson-Urquhart S, Schuh S, Sherman PM, Farion KJ, Gouin S, Willan AR, Goeree R, Johnson DW, Black K, Schnadower D, Gorelick MH; Pediatric Emergency Research Canada (PERC) Gastroenteritis Study Group. Impact of emergency department probiotic treatment of pediatric gastroenteritis: study protocol for the PROGUT (Probiotic Regimen for Outpatient Gastroenteritis Utility of Treatment) randomized controlled trial. Trials. 2014 May 14;15:170. doi: 10.1186/1745-6215-15-170. PMID 24885220

RESULTS

PARTICIPANT FLOW:
Groups:
- Lactobacillus Rhamnosus GG: LGG 10^10 cfu PO bid x 5 days
  LGG: LGG 10^10 cfu PO BID X 5 days
Period: Overall Study
Arm/Group | Lactobacillus Rhamnosus GG | Placebo
Started | 483 | 488
Completed | 468 | 475
Not Completed | 15 | 13
Not completed — Lost to Follow-up | 15 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactobacillus Rhamnosus GG | Placebo | Total
Number analyzed (Participants) | 483 | 488 | 971
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 1.4 [0.9 to 2.4] | 1.4 [0.8 to 2.3] | 1.4 [0.9 to 2.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 236 | 222 | 458
  Male | 247 | 266 | 513
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 0 | 9
  Asian | 8 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 176 | 162 | 338
  White | 144 | 163 | 307
  More than one race | 24 | 16 | 40
  Unknown or Not Reported | 121 | 138 | 259
Region of Enrollment [Number; unit: participants]
  United States | 483 | 488 | 971
Median Modified Vesikari Scale score at presentation [Median (Inter-Quartile Range); unit: units on a scale] — The modified Vesikari scale is a validated global gastroenteritis severity scale that includes duration and severity of vomiting and diarrhea, maximum recorded temperature, unscheduled health care visits and types of treatment received. Scores range from 0 to 20, with higher scores indicating more severe disease). A score of 9 or greater is considred moderate to severe gastroenteritis
  units on a scale | 12 [10 to 14] | 12 [9 to 14] | 12 [10 to 14]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Modified Vesikari Scale Score >=9
Description: This is a validated gastroenteritis severity score that includes duration and frequency of diarrhea, duration and frequency of vomiting, duration and frequency of fever and use of health care resources. Scores >=9 indicate moderate-severe gastroenteritis. Higher is worse.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lactobacillus Rhamnosus GG | Placebo
Number analyzed (Participants) | 468 | 475
Participants | 55 | 60
Statistical Analysis 1: Comparison: Lactobacillus Rhamnosus GG vs Placebo; Test type: Superiority; p = 0.83, Mantel Haenszel

2. Secondary Outcome: Number of Participants With LGG Bacteremia
Description: bacteremia caused by LGG
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Lactobacillus Rhamnosus GG | Placebo
Number analyzed (Participants) | 468 | 475
Participants | 0 | 0

3. Secondary Outcome: Diarrhea Duration
Description: diarrhea duration in hours after randomization
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Lactobacillus Rhamnosus GG | Placebo
Number analyzed (Participants) | 468 | 475
hours | 49.7 [18.8 to 86.4] | 50.9 [25.0 to 88.2]
Statistical Analysis 1: Comparison: Lactobacillus Rhamnosus GG vs Placebo; Test type: Superiority; p = 0.26, Van Elteren's modification Mann-Whitney

ADVERSE EVENTS:
Time Frame: 35 days, long term follow up 1 year
Arm/Group | Lactobacillus Rhamnosus GG | Placebo
All-Cause Mortality (participants affected / at risk) | 0/483 | 0/488
Serious Adverse Events (participants affected / at risk) | 8/483 | 13/488
Other Adverse Events (participants affected / at risk) | 55/483 | 49/488
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lactobacillus Rhamnosus GG (N=483) | Placebo (N=488)
Worsening diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (4)
ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
seizure (Nervous system disorders) | 1 (1) | 1 (1) — febrile
lethargy (Nervous system disorders) | 1 (1) | 1 (1)
lower respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
dehydration (Gastrointestinal disorders) | 1 (1) | 2 (2)
metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
fever (General disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lactobacillus Rhamnosus GG (N=483) | Placebo (N=488)
other (Gastrointestinal disorders) | 40 (40) | 35 (35)
other (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT01773967/Prot_SAP_000.pdf